CLINICAL TRIAL: NCT01339988
Title: Treatment Plan for Hematologic Malignancies Using Intravenous Busulfan and Cyclophosphamide Instead of Total Boby Irradiation (TBI) and Cyclophosphamide to Examine Results, Success and Side Effects of Treatment With Chemotherapy Only, as a Preparative Therapy for Patients With Cord Blood Transplants
Brief Title: Busulfan and Cyclophosphamide Instead of Total Boby Irradiation (TBI) and Cyclophosphamide for Hematological Malignancies Hematocrit (HCT)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Menachem Bitan, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-11-MB-442-CTIL
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Acute Leukemias; Chronic Leukemias; Myelodysplastic Syndrome; Juvenile Myelomonocytic Leukemia
Keywords: Stem-cells; Transplantation; Busulfex; Cyclophosphamide; Total-Body-Ittadiation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile | interventions — Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busulfan/Cyclophosphamide (Experimental)
  Interventions: Drug: Busulfan/Cyclophosphamide

INTERVENTIONS:
Drug: Busulfan/Cyclophosphamide — Conditioning regimen:
  Cyclophosphamide 50mg/kg/day for 4 days + Busulfan 0.8-1.0mg/kg/day for 4 days.
  Other Names: Cytoxan

SUMMARY:
Long-term follow-up studies have demonstrated significant late toxicities of total body irradiation (TBI), which are most marked in children radiated at a young age. Growth failure, decline in cognitive function, and endocrine abnormalities have all been described. Good outcomes can be achieved with alkylating agents only as a preparative regimen. This plan will use a combination of busulfan and cyclophosphamide (Bu/Cy) with or without antithymocyte globulin (ATG) to reduce the late toxicities of therapy that includes TBI.

ELIGIBILITY:
Inclusion Criteria:

* Suitable cord blood from matched unrelated or related donor.
* Cardiac (Echo/EKG): shortening fraction ≥ 27%
* Electrolytes within normal CCHMC limits.
* Pulmonary function tests: DLCO ≥ 50%
* Renal: creatinine clearance/GFR ≥ 60 ml/minute/1.73m2
* Lumbar puncture: no leukemic infiltrate.
* CBC: ANC ≥ 1000ml and unsupported platelet count of ≥ 50,000/ml
* Documented HSV and CMV titers, Hepatitis B surface antigen, Hepatitis C by serology, HIV by serology: all negative.
* Hepatic transaminases < 2.5x normal; Total bilirubin < 2 mg/dl Patients who do not meet above organ function criteria (liver, cardiac, renal), due to the presence of a tumor compromising these organs, may have exception made for these criteria and remain eligible for treatment plan after consultation with Program Director of Blood and Marrow Transplant

Exclusion Criteria:

* Patients with neoplastic or non-neoplastic disease of any major organ system that would compromise their ability to withstand the pre-transplant conditioning regimen.
* Patients with uncontrolled (culture or biopsy positive) infections requiring intravenous antivirals, antibiotics, or antifungals. Patients on prolonged antifungal therapy with a history of fungal infection should be considered for a non-myeloablative protocol.
* Patients who are pregnant or lactating. Patients of childbearing potential must practice an effective method of birth control while participating on this treatment plan.
* HIV seropositive patients

Max Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Five years

SECONDARY OUTCOMES:
Disease free survival | Five years